CLINICAL TRIAL: NCT05784896
Title: Predictors Of Chronic Thromboembolic Pulmonary Hypertension Following Acute Pulmonary Embolism
Brief Title: CTEPH Predictors Following Acute Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Abd Elhamied, Assistant lecturer, Assiut University
Other Study IDs: CTEPH predictors in acute PE
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: CTEPH Predictors
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: v/Q scanning & CT pulmonary angiography & Echocardiography — Echocardiography ( comparative follow up of the RVSF PASP TAPSE IVC).
  CT pulmonary angiography with assessment of the following parameters :
  Intravascular web. dilated bronchail arteries. Arterial retraction. dilated pulmonary arteries. RV/LV diameter more than 1. Flattening of interventricular septum. V/Q scanning Following ESC/ERS Guideline recommendations, V/Q is the preferred and recommended test for CTEPH. It has a sensitivity of >96% and normal V/Q scan can rule out CTEPH . V/Q lung scintigraphy was interpreted as positive for CTEPH if there was at least one segmental or two sub-segmental mismatched perfusion defects, as proposed by the European Association of Nuclear Medicine (EANM) guidelines for the diagnosis of acute PE.

SUMMARY:
Identify risk factors for developing chronic thromboembolic pulmonary hypertension after acute pulmonary embolism.

Determine echocardiographic predictors of chronic thromboembolic pulmonary hypertension.

Determine the radiological predictors of chronic thromboembolic pulmonary hypertension in CT pulmonary angiography.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension(CTEPH) is considered to be a long-term complication after acute pulmonary embolism (PE) characterized by persistent perfusion defects of pulmonary arteries caused by fibrotic remodeling. Its pathophysiology has not been fully elucidated yet, although it has been accepted that the increased pulmonary vascular resistance is caused by obstruction of pulmonary arterial vessels by organized thromboemboli and by vascular remodeling of small un obstructed vessels. (1) Although CTEPH had been thought to develop in relatively few patients post-pulmonary thromboembolism, the latest data suggest an unexpectedly high incidence of approximately 4%. (2) In addition, although there are well-defined risk factors for pulmonary thromboembolism, the risk factors for CTEPH have not yet been sufficiently defined. (3) For that reason, the determination of risk factors is of great importance for the early diagnosis of patients with CTEPH, with its high mortality and morbidity. The clinical presentation of CTEPH is characterized by non-specific symptoms and include exercise intolerance, dyspnea, fatigue, chest pain, and syncope (at exercise). These symptoms are also consistent with other more common cardiopulmonary conditions such as asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease, coronary artery disease, cardiac arrhythmia or heart failure not caused by chronic pulmonary thrombi. (4) These non-specific symptoms are commonly reported by patients who suffered from an acute PE and therefore, the possibility of CTEPH can be frequently considered . The diagnostic management of CTEPH is complex. In many patients pulmonary perfusion scintigraphy, transthoracic echocardiography and conventional pulmonary angiography with determination of pulmonary hemodynamics need to be performed before the diagnosis of CTEPH can be refuted. (5)

ELIGIBILITY:
Inclusion Criteria:

All adult patients of both gender more than 18 yrs admitted at chest department and diagnosed by CT pulmonary angiography as acute pulmonary embolism during a period of one year will be recruited in the study.

About 80 patients as the average number of patients admitted per month is 7.

Exclusion Criteria:

Patients with congenital or acquired heart diseases. Patients with chronic chest diseases. Patients previously diagnosed chronic thromboembolic pulmonary hypertension by V/Q scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients of both gender more than 18 yrs admitted at chest department and diagnosed by CT pulmonary angiography as acute pulmonary embolism during a period of one year will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Identify risk factors for devolping chronic thromboembolic pulmonary hypertention after acute pulmonary embolism. | baseline
  Follow up to patients with acute pulmonary embolism after 3 months with V/Q scanning and ECHO

REFERENCES:
- [Background] Klok FA, Dzikowska-Diduch O, Kostrubiec M, Vliegen HW, Pruszczyk P, Hasenfuss G, Huisman MV, Konstantinides S, Lankeit M. Derivation of a clinical prediction score for chronic thromboembolic pulmonary hypertension after acute pulmonary embolism. J Thromb Haemost. 2016 Jan;14(1):121-8. doi: 10.1111/jth.13175. Epub 2015 Dec 29. PMID 26509468
- [Background] Dentali F, Donadini M, Gianni M, Bertolini A, Squizzato A, Venco A, Ageno W. Incidence of chronic pulmonary hypertension in patients with previous pulmonary embolism. Thromb Res. 2009 Jul;124(3):256-8. doi: 10.1016/j.thromres.2009.01.003. Epub 2009 Feb 3. PMID 19193397
- [Background] Auger WR, Kim NH, Kerr KM, Test VJ, Fedullo PF. Chronic thromboembolic pulmonary hypertension. Clin Chest Med. 2007 Mar;28(1):255-69, x. doi: 10.1016/j.ccm.2006.11.009. PMID 17338940
- [Background] Dyspnea. Mechanisms, assessment, and management: a consensus statement. American Thoracic Society. Am J Respir Crit Care Med. 1999 Jan;159(1):321-40. doi: 10.1164/ajrccm.159.1.ats898. No abstract available. PMID 9872857
- [Background] Klok FA, Surie S, Kempf T, Eikenboom J, van Straalen JP, van Kralingen KW, van Dijk AP, Vliegen HW, Bresser P, Wollert KC, Huisman MV. A simple non-invasive diagnostic algorithm for ruling out chronic thromboembolic pulmonary hypertension in patients after acute pulmonary embolism. Thromb Res. 2011 Jul;128(1):21-6. doi: 10.1016/j.thromres.2011.03.004. Epub 2011 Mar 30. PMID 21450333
- [Background] Bova C, Vanni S, Prandoni P, Morello F, Dentali F, Bernardi E, Mumoli N, Bucherini E, Barbar S, Picariello C, Enea I, Pesavento R, Bottino F, Jimenez D; Bova Score Validation Study Investigators. A prospective validation of the Bova score in normotensive patients with acute pulmonary embolism. Thromb Res. 2018 May;165:107-111. doi: 10.1016/j.thromres.2018.04.002. Epub 2018 Apr 4. PMID 29631073